CLINICAL TRIAL: NCT02494401
Title: Taking Charge of Systemic Sclerosis: Improving Patient Outcomes Through Self-management
Brief Title: Taking Charge of Systemic Sclerosis
Acronym: TOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of New Mexico (Other); Medical University of South Carolina (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Dinesh Khanna, MD, MS, Dinesh Khanna, MD,MS, PI, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CER-1310-08323.
Record Dates: First submitted 2015-05-22; First posted 2015-07-10 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Scleroderma
Keywords: systemic sclerosis; ssc
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based self-management program (Active Comparator): Internet-based self-management program Patients randomized to active treatment intervention will be assigned to the Internet program. The site will be accessed via secured website. The modules will be presented 1-2 per week and will be moderated by a researcher with expertise in moderating Discussion Boards.
  Interventions: Other: Internet-based self-management program
- Education book group (Other): Educational book group. Participants in the control group will receive a copy of The Scleroderma Book: A Guide for Patients and Families, by Dr. Maureen Mayes.
  Interventions: Other: Scleroderma book

INTERVENTIONS:
Other: Internet-based self-management program
  Arms: Internet-based self-management program
Other: Scleroderma book
  Arms: Education book group

SUMMARY:
This Study is a collaborative project with partners (people with scleroderma and stakeholders) designed to refine an internet program for patients with scleroderma and to compare the internet program to an authoritative educational book (Taking Charge of Systemic Sclerosis [TOSS]). During a 16-week comparative effectiveness 16-week randomized controlled trial, the investigators will recruit up to 250 patients who will be randomized to either TOSS or authoritative book for patients, The Scleroderma Book: A Guide for Patients and Families.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be residents of the United States
* Diagnosed with systemic scleroderma,
* 18 years of age
* Possess basic computer literacy and have access to a computer with Internet and email capabilities
* Have the ability to communicate in English

Exclusion Criteria:

* No computer access
* Inability to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2016-03-06 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Poole, Principal Investigator — University of New Mexico; Dinesh Khanna, Principal Investigator — University of Michigan; Richard Silver, Principal Investigator — Medical University of South Carolina
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Murphy SL, Whibley D, Kratz AL, Poole JL, Khanna D. Fatigue Predicts Future Reduced Social Participation, not Reduced Physical Function or Quality of Life in People with Systemic Sclerosis. J Scleroderma Relat Disord. 2021 Jun 1;6(2):187-193. doi: 10.1177/2397198320965383. Epub 2020 Sep 20. PMID 34337153
- [Derived] Khanna D, Serrano J, Berrocal VJ, Silver RM, Cuencas P, Newbill SL, Battyany J, Maxwell C, Alore M, Dyas L, Riggs R, Connolly K, Kellner S, Fisher JJ, Bush E, Sachdeva A, Evnin L, Raisch DW, Poole JL. Randomized Controlled Trial to Evaluate an Internet-Based Self-Management Program in Systemic Sclerosis. Arthritis Care Res (Hoboken). 2019 Mar;71(3):435-447. doi: 10.1002/acr.23595. Epub 2019 Feb 5. PMID 29741230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment occurred at two sites, The University of Michigan and the Medical University of South Carolina. Recruitment also took place utilizing social media, with the help of our patient partners and the Sclerderma Foundation and Scleroderma Research Foundation.
Pre-assignment Details: Participants completed baseline questionnaires. Participants were randomized to the intervention or control condition using a 1:1 ratio and computer-generated block randomization, and were stratified based on scores on the Patient Health Questionnaire-8 (<10, >10) in the baseline questionnaire.
Groups:
- Internet-based Self-management Program: Internet-based self-management program Patients randomized to active treatment intervention will be assigned to the Internet program. The site will be accessed via secured website. The modules will be presented 1-2 per week and will be moderated by a researcher with expertise in moderating Discussion Boards.
  Internet-based self-management program
- Education Book Group: Educational book group. Participants in the control group will receive a copy of The Scleroderma Book: A Guide for Patients and Families, by Dr. Maureen Mayes.
  Scleroderma book
Period: Overall Study
Arm/Group | Internet-based Self-management Program | Education Book Group
Started | 134 | 133
Week 16 | 123 | 124
6 Month Follow up | 109 | 106
Completed | 109 | 106
Not Completed | 25 | 27
Not completed — Lost to Follow-up | 22 | 25
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet-based Self-management Program | Education Book Group | Total
Number analyzed (Participants) | 134 | 133 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] — age at time of enrollment
  years | 54.3 (10.1) | 52.9 (13.1) | 53.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 120 | 243
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 105 | 102 | 207
  Unknown or Not Reported | 22 | 27 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 7 | 13 | 20
  White | 112 | 109 | 221
  More than one race | 11 | 5 | 16
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 134 | 133 | 267
Managing Symptoms Scale on the PROMIS® Self-efficacy Short Form 8 [Mean (Standard Deviation); unit: T-Score] — Managing Symptoms score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident). The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage symptoms.
  T-Score | 47.41 (9.15) | 47.58 (7.81) | 47.50 (8.49)
Quality of Life on the European Quality of Life-5 Dimensions (EQ-5D) Scale [Mean (Standard Deviation); unit: units on a scale] — The (EQ-5D) provides a generic health-related quality of life assessment. The 5 domains listed in each row are scored into 3 levels, level 1 (no problem), level 2 (some problems), level 3 (extreme problems).
  Visual analogue scale is a vertical scale with end points of 0 and 100, 0 corresponds to " the worst health you can imagine", and 100 corresponds to "the best health you can imagine".
  Using a conversion algorithm, the EQ-5D index patient responses are converted into a health utility measure, ranging from 0.0 (death) to 1.0 (full or optimal health).
  units on a scale
    Mobility | 1.53 (0.52) | 1.61 (0.49) | 1.57 (0.50)
    Self-Care | 1.28 (0.48) | 1.79 (0.49) | 1.31 (0.49)
    Usual Activities | 1.78 (0.50) | 1.79 (0.43) | 1.79 (0.46)
    Pain Discomfort | 1.93 (0.48) | 2.02 (0.43) | 1.98 (0.46)
    Anxiety | 1.56 (0.61) | 1.63 (0.62) | 1.60 (0.61)
    Visual Analogue Scale | 67.47 (18.01) | 63.72 (17.33) | 65.6 (17.74)
    EQ-5D Index | 0.71 (0.18) | 0.69 (0.16) | 0.70 (0.17)
Confidence in Self Management on the Patient Activation Measure Scale [Count of Participants; unit: Participants] — The Patient Activation Measure (PAM) is a 13-item measure that assesses patient knowledge, skill, and confidence for self-management.PAM scores were categorized into 4 levels: level 1, the individual is disengaged/overwhelmed; level 2, the individual is aware but struggling; level 3, the individual is taking action;and level 4, the individual is maintaining behavior.The summed score is finally transformed into a 0-100 point scale with higher scores indicating more confidence and knowledge in patients managing their condition
  Participants
    Patient Activation Level 1 | 14 | 14 | 28
    Patient Activation Level 2 | 15 | 15 | 30
    Patient Activation Level 3 | 23 | 27 | 50
    Patient Activation Level 4 | 82 | 77 | 159
Appearance Satisfaction on the Satisfaction With Appearance Scale (SWAP) Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Satisfaction with Appearance Scale (SWAP) is a 6-item scale measuring body image concerns and social discomfort with body parts. It is scored from 0 to 36, with higher scores associated with greater dissatisfaction.
  units on a scale | 17.1 (9.53) | 16.81 (8.13) | 16.96 (8.85)
Managing Daily Activities Scale on the PROMIS® Self-efficacy Short Form 8 [Mean (Standard Deviation); unit: T-score] — Managing Daily Activities score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage daily actvities.
  T-score | 44.83 (7.60) | 44.71 (6.77) | 44.77 (7.19)
Managing Emotions Scale on the PROMIS® Self-efficacy Short Form 8 [ [Mean (Standard Deviation); unit: T-Score] — Managing Emotions score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident) this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage emotions.
  T-Score | 46.78 (9.29) | 46.34 (8.75) | 46.56 (9.01)
Managing Medications and Treatment Scale on the PROMIS® Self-efficacy Short Form 8 [Mean (Standard Deviation); unit: T-Score] — Managing Medication and Treatment score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident) this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage medications and treatments.
  T-Score | 49.15 (9.06) | 50.3 (8.29) | 49.72 (8.69)
Managing Social Interactions Scale on the PROMIS® Self-efficacy Short Form 8 [Mean (Standard Deviation); unit: T Score] — Managing Social Interactions score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident) this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage social interactions.
  T Score | 46.57 (9.74) | 46.66 (8.96) | 46.62 (9.34)
Physical Function scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T Score] — Physical Function domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10.A higher score represents better physical function, a lower score represents poorer physical function.
  T Score | 40.63 (6.95) | 40.17 (6.15) | 40.4 (6.95)
Social Role scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T Score] — Social role domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
  T Score | 43.74 (8.63) | 44.39 (7.68) | 44.06 (8.17)
Anxiety scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T Score] — Anxiety domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much),this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
  T Score | 53.85 (9.72) | 54.11 (10.31) | 53.98 (10.0)
Depression scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T-Score] — Depression domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much),this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
  T-Score | 51.04 (10.03) | 51.59 (9.69) | 51.31 (9.85)
Fatigue scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T-Score] — Fatigue domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much),this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
  T-Score | 58.47 (10.52) | 58.91 (10.31) | 58.69 (10.40)
Pain Interference scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T-Score] — Pain interference domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much). A raw score is created from each short form that makes up the Profile. To find the total raw score for a short form with all questions answered, sum the values of the response to each question within each domain. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
  T-Score | 57.99 (9.37) | 57.92 (9.22) | 57.95 (9.28)
Visual Analogue Scale Pain Intensity scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T Score] — the visual analogue scale pain intensity in the PROMIS-29 Profile v2.0® are scored as 0 being no pain and 10 being the worst imaginable pain.
  T Score | 4.08 (2.21) | 4.25 (2.26) | 4.16 (2.24)
Sleep Disturbance scale on the PROMIS® 29 Profile v 2.0 outcome measure [Mean (Standard Deviation); unit: T-score] — Sleep disturbance domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much),this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
  T-score | 55.22 (6.96) | 56.18 (7.84) | 55.7 (7.41)
PHQ-8 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-8 (PHQ-8) is an 8-item questionnaire that is commonly used to measure depressive symptoms. The minimum score is 0 with a maximum score of 24. A score of ≥10 is consistent with depressed mood, a score of ≥20 is consistent with severely depressed mood.
  units on a scale | 8.61 (5.39) | 8.72 (4.98) | 8.67 (5.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in Managing Symptoms Scale on the PROMIS® Self-efficacy Short Form 8
Description: Managing Symptoms score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage symptoms.
Time Frame: Baseline compared with 16 weeks, 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.35 (6.12) | 0.94 (6.79)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.50 (7.13) | 1.49 (6.67)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney) — p value for 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney) — p value for 6 month comparison

2. Secondary Outcome: Change in Quality of Life on the European Quality of Life-5 Dimensions (EQ-5D) Index Scale
Description: EQ-5D index scale uses a conversion algorithm to convert the raw scores into a health utility measure, ranging from 0.0 (death) to 1.0 (full or optimal health).
Time Frame: Baseline compared with 16 weeks, 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.002 (0.14) | 0.02 (0.14)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.002 (0.12) | 0.04 (0.15)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — p value 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney) — p value 6 month comparison

3. Secondary Outcome: Change in Confidence in Self Management on the Patient Activation Measure Scale
Description: The Patient Activation Measure (PAM) is a 13-item measure that assesses patient knowledge, skill, and confidence for self-management. Each item is scored from 1 (strongly disagree) to 4 (strongly agree). PAM scores were categorized into 4 levels: level 1, the individual is disengaged/overwhelmed; level 2, the individual is aware but struggling; level 3, the individual is taking action;and level 4, the individual is maintaining behavior. The analysis will look at any change in these levels where level 4 denotes someone as full "activated".
Time Frame: Baseline compared with 16 weeks, 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: PAM level
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
PAM level
  16 weeks | 0.83 (4.98) | 0.98 (5.55)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.90 (5.22) | 1.70 (4.50)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — p value baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Brief Satisfaction on the Satisfaction With Appearance Scale (SWAP) Scale
Description: The Brief Satisfaction with Appearance Scale (SWAP) is a 6-item scale measuring body image concerns and social discomfort with body parts. It is scored from 0 to 36, with higher scores associated with greater dissatisfaction.
Time Frame: Baseline compared with 16 weeks, 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.82 (10.58) | 0.31 (9.56)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.18 (10.19) | 0.91 (9.88)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

5. Secondary Outcome: Change in Managing Daily Activities Scale on the PROMIS® Self-efficacy Short Form 8
Description: Managing Daily Activities score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage symptoms.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.17 (5.11) | 0.79 (4.52)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.04 (4.56) | 0.48 (6.28)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — p value baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney) — p value for 6 month comparison

6. Secondary Outcome: Change in Managing Emotions Scale on the PROMIS® Self-efficacy Short Form 8
Description: Managing Emotions score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage symptoms.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.09 (6.28) | 0.73 (5.34)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.71 (7.61) | 1.22 (7.66)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney) — p value for baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney) — p value for 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney) — p value for 6 month comparison

7. Secondary Outcome: Change in Managing Medications and Treatment Scale on the PROMIS® Self-efficacy Short Form 8
Description: Managing Medication and Treatment score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage symptoms.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.54 (7.59) | 0.70 (6.29)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.89 (8.31) | 0.49 (8.50)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney) — p value for baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney) — p value for 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney) — p value for 6 month comparison

8. Secondary Outcome: Change in Managing Social Interactions Scale on the PROMIS® Self-efficacy Short Form 8
Description: Managing Social Interactions score on the PROMIS® Self-efficacy Short Form 8 consists of 8 items scored from 1 (not at all confident) to 5 (very confident), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. Higher scores are indicative of greater ability to manage symptoms.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.43 (6.94) | 0.99 (7.42)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.40 (8.12) | 1.47 (7.95)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.93, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

9. Secondary Outcome: Change in Physical Function Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: Physical Function domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents better physical function, a lower score represents poorer physical function.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.05 (5.71) | 0.75 (4.83)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.09 (4.93) | 1.08 (5.84)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

10. Secondary Outcome: Change in Social Role Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: Social role domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents better social role functioning and a lower score represents poorer social role functioning.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 2.05 (17.19) | 2.24 (15.58)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 1.19 (17.15) | 1.65 (15.29)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.93, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.84, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

11. Secondary Outcome: Change in Anxiety Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: Anxiety domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.16 (6.93) | 0.86 (7.64)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.40 (8.55) | -1.14 (8.35)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

12. Secondary Outcome: Change in Depression Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: Depression domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.08 (6.40) | 0.13 (6.76)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.61 (7.75) | -1.23 (7.95)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

13. Secondary Outcome: Change in Fatigue Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: Fatigue domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.005 (6.90) | 0.20 (7.19)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | 0.78 (6.90) | -1.36 (8.36)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

14. Secondary Outcome: Change Pain Interference Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: Pain interference domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much), this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | -0.65 (6.96) | -0.80 (6.95)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | -0.58 (7.29) | -1.03 (8.84)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

15. Secondary Outcome: Change in Visual Analogue Scale Pain Intensity Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: The visual analogue scale pain intensity in the PROMIS-29 Profile v2.0® is scored as 0 being no pain and 10 being the worst imaginable pain.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | 0.11 (1.78) | 0.19 (1.78)
  6 months: number analyzed (Participants) | 109 | 107
  6 months | 0.02 (1.91) | -0.09 (2.32)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.7, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

16. Secondary Outcome: Change in Sleep Disturbance Scale on the PROMIS® 29 Profile v 2.0 Outcome Measure
Description: Sleep disturbance domain in the PROMIS-29 Profile v2.0® are scored from 1 (unable to do/never/not at all) to 5 (without any difficulty/always/very much),this provides a raw score. The raw score is translated to a T-Score using a conversion table supplied by the Assessment Center. A score of 50 is the average for the US general population with a standard deviation of 10. A higher score represents worse symptomatology, a lower score represents better symptomatology.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | -2.95 (6.22) | -3.40 (6.62)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | -1.30 (6.74) | -1.92 (6.65)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

17. Other Pre Specified Outcome: Change in PHQ-8
Description: The Patient Health Questionnaire-8 (PHQ-8) is an 8-item questionnaire that is commonly used to measure depressive symptoms. A score of ≥10 is consistent with depressed mood with a score ranging from 0 to 24.
Time Frame: Baseline compared to 16 weeks and 6 months
Population: Population analyzed at 6 months differs due to drop outs shown in participant flow table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based Self-management Program | Education Book Group
Number analyzed (Participants) | 123 | 124
units on a scale
  16 weeks | -1.19 (5.02) | -1.27 (4.99)
  6 months: number analyzed (Participants) | 109 | 106
  6 months | -1.79 (5.06) | 1.63 (5.12)
Statistical Analysis 1: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney) — p value of baseline comparison
Statistical Analysis 2: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — p value of 16 week comparison
Statistical Analysis 3: Comparison: Internet-based Self-management Program vs Education Book Group; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney) — p value of 6 month comparison

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Internet-based Self-management Program | Education Book Group
All-Cause Mortality (participants affected / at risk) | 1/134 | 0/133
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/133
Other Adverse Events (participants affected / at risk) | 0/134 | 0/133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT02494401/Prot_SAP_000.pdf